CLINICAL TRIAL: NCT02634398
Title: A Post Market ObServational StudY on the Effect of DRG StiMulation in PATients witH Chronic Pain Following Surgical Lumbar DiscectomY (Failed Back Surgery Syndrome): SYMPATHY
Brief Title: A Post Market Study on DRG Stimulation in FBSS (SYMPATHY)
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollments
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 26-SMI-2015
Record Dates: First submitted 2015-10-23; First posted 2015-12-18 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated subjects: All subjects recruited and treated wiht the Axium neurostimulator

SUMMARY:
The purpose of this Post Market Observational Study is to monitor the effect of the Axium® SCS System in the management of chronic pain following surgical lumbar discectomy in subjects whom are routinely scheduled for treatment with the Axium® SCS System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic pain following surgical lumbar discectomy for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the VAS in the subjects' primary area of pain
6. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
5. Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects with indwelling devices that may pose an increased risk of infection
8. Subjects currently has an active infection
9. Subject has participated in another clinical investigation within 30 days
10. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
11. Subject has been diagnosed with cancer in the past 2 years.
12. Subject has an anatomical spinal abnormality which is anticipated to require further surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic pain post discectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain Relief | Post implantation at; 1 week and 1, 3, 6 and 12 months
  Assessed by change in pain intensity on a Visual Analogue Scale (VAS) from pre-treatment baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Antalgie de l'EHC-Hôpital de Morges, Morges, Canton of Vaud, Switzerland